CLINICAL TRIAL: NCT07115134
Title: Efficacy of a Novel Prototype Gastrostomy Tube Anchor Dressing
Acronym: Tube Anchor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001158
Record Dates: First submitted 2025-07-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gastroenterology Surgery; Tube Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Bearables Gastrostomy Tube Dressing Prototype (Experimental)
  Interventions: Device: Bearables Gastrostomy Tube Dressing

INTERVENTIONS:
Device: Bearables Gastrostomy Tube Dressing — The gastrostomy tube dressing in its current design is composed of two parts, both of which are external to the patient: one part is rigid and holds the gastrostomy at a fixed position, this is a 3D printed design that is produced here. The second part is a 3" x 3" flexible, cushioned, biocompatible adhesive bandage designed to fit around the skin opening (Silicone Foam Dressing, NH NeuHeils, USA). The design is subject to minor changes including the number of parts and location with the structure of the padding and securement but will continue to be designed with comfort as a priority. After assembly, the device is packaged (sterilization pouches, Plastcareusa, USA), sealed, and sanitized using UV light prior to patient use.

SUMMARY:
This is a single-center prospective study evaluating the efficacy of a prototype gastrostomy anchor dressing for use with button gastrostomy tubes. The anchor dressing has been previously evaluated for usability by parents, patients, and nurses. This study compares several outcomes related to complications from gastrostomy tube placement using a prospective cohort of patients and a retrospective analysis of complications associated with gastrostomy tubes. Prospective patients will initially be monitored until they have completed their last dressing change or for a maximum of 50 days. They will then complete their final survey. Their charts will be reviewed for up to one year from their initial gastrostomy placement. The study's primary objective is to determine if the novel gastrostomy tube anchor dressing reduces rates of gastrostomy tube dislodgement and ED/clinic visits for gastrostomy tube complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing gastrostomy tube placement or are within five days post-operatively of gastrostomy tube placement.

Exclusion Criteria:

* 1. Patients with a skin condition that limits the placement of the dressing, this will be confirmed with the clinical team

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Rates Gastrostomy Tube Dislodgement Before and After Dressing Placement | Up to one year
  Current rates of gastrostomy tube complications and dislodgement will be evaluated with our retrospective review, then compared to rates of complications and dislodgement after our novel dressing placement. This was chosen as complications after gastrostomy tube placement are high, and we believe that our dressing will lower them.
Gastrostomy tube complications | Up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No